CLINICAL TRIAL: NCT00001198
Title: Biochemical, Physiological, and Psychological Measures in Normal Controls and Relatives of Psychiatric Patients
Brief Title: Evaluating Genetic Risk Factors for Childhood-Onset Schizophrenia
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 840050; 84-M-0050
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10-10

CONDITIONS: Psychosis; Schizophrenia; Genetic Structure; Childhood Onset Psychotic Disorders; Schizoaffective Disorder
Keywords: Schizophrenia; Observational
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

SUMMARY:
A study of children and adolescents (current N=100) with very early onset by age 12 (COS) of DSM-III-R defined schizophrenia with (97-M-0126) is examining the clinical, neurobiological, early neurodevelopmental, genetic, and clinical drug response characteristics of these cases. Earlier studies have documented the continuity between COS and adult onset cases (See Jacobsen and Rapoport, 1998 for review). The focus has now shifted to increasing the sample size and evaluation of familial risk factors including: psychiatric diagnoses of family members; smooth pursuit eye movements; neuropsychological tests deficits, and obtaining blood for cell lines for genetic studies (family members only, this is also covered under 96-M-0060, Dr. Ellen Sidransky).

A study of obstetrical records of COS probands indicated no increase in adverse pre or perinatal events for these cases compared with obstetrical records of their siblings (Nicolson et al submitted). In contrast, several findings point to increased risk for these probands. To date, a total of 5 (10.4%) COS subjects were found to have previously unknown cytogenetic abnormalities (Microdeletion of 22q11 (3 cases), (Usiskin et al, submitted), Mosaic 45X0 (one case) (Kumra et al, 1998) and balanced 1:7 translocation (Gordon et al 1994).

The study of first degree relatives of these very rare cases addresses the hypothesis that risk factors, most probably genetic, are increased in immediate family members relative both to community controls and to the relatives of patients with chronic, treatment resistant, adult-onset schizophrenia (AOS). A second hypothesis is that COS familial risk factors show significant relationship to the developmental delays/abnormalities being observed in the COS probands. As a total of 50 additional COS subjects will be studied over the next 5 years, the pediatric control sample for the probands will also be increased, determined by the need to have concurrent measures for patients and controls to maintain measurement validity. Thus a total of 600 additional subjects are to be studied including 50 controls for COS probands, 150 COS relatives, 150 controls for COS relatives, and 250 relatives of adult onset schizophrenics (AOS).

DETAILED DESCRIPTION:
A study of children and adolescents with very early onset by age 12 (COS) of DSM-III-R defined schizophrenia is examining the clinical, neurobiological, early neurodevelopmental, genetic, and clinical drug response characteristics of these cases, under Protocols 97-M-0126 and 03-M-0035. Earlier studies have documented the continuity between COS and adult-onset cases. The focus has now shifted to increasing the sample size and evaluation of familial risk factors including: psychiatric diagnoses of family members; neuropsychological testing, anatomic and functional brain imaging, and obtaining blood and fibroblasts for cell lines for genetic studies.

A study of obstetrical records of COS probands indicated no increase in adverse pre or perinatal events for these cases compared with obstetrical records of their well siblings. In contrast, several findings point to increased genetic risk for these probands.

The study of first-degree relatives of these very rare cases addresses the hypothesis that risk factors, most probably genetic, are increased in immediate family members relative both to community controls and to the relatives of patients with chronic, treatment resistant, adult-onset schizophrenia (AOS). A second hypothesis is that COS familial risk factors include similar forms of the developmental delays/abnormalities being observed in the COS probands. Preliminary data suggests greater abnormalities of frontal-parietal circuits for early onset patients and their relatives than seen in adult onset illness.

We will examine brain development in unrelated healthy volunteers and siblings of our COS probands by combining resting- and task-related magnetic resonance imaging (MRI) and magnetoencephalography (MEG) imaging. Imaging studies may lead to greater understanding of the course, mechanisms, and influences on brain development of high-risk siblings and may lead to improved understanding of the risk factors, early identification, and optimization of brain maturation. For more than 20 years, imaging has been done under a separate protocol (89-M-0006); however, we now plan to incorporate these imaging studies into this protocol (as well as into our main patient screening and follow-up protocol (03-M-0035) by previously submitted amendment).

ELIGIBILITY:
* INCLUSION CRITERIA:

  i. For Healthy Controls
* Age 6 and above
* Evidence of normal developmental history and normal functioning

ii. For Relatives of Probands

* Ages 6 and above
* Evidence of blood relationship to proband with a disorder under study, with usual selection of first-degree relatives, and occasional participation of more distantly-related relatives (e.g., grandparents, aunts/uncles, cousins).

EXCLUSION CRITERIA :

i.For Healthy Controls

* Evidence of medical or neurological disease
* Diagnosis of schizophrenia or schizoaffective disorder or in first-degree relatives by history, clinical interview, or by structured, diagnostic psychiatric interview (Diagnostic Interview for Children and Adolescents -IV)

ii.For Relatives of Probands

* Absence of consent on the part of the proband or parent(s) of proband to contact relatives
* Absence of signed consent or assent by relative(s) to participate
* Lack of consent capacity

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1556 (Actual)
Dates: Start 1984-03-19; Study Completion 2017-10-10

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Casey BJ, Castellanos FX, Giedd JN, Marsh WL, Hamburger SD, Schubert AB, Vauss YC, Vaituzis AC, Dickstein DP, Sarfatti SE, Rapoport JL. Implication of right frontostriatal circuitry in response inhibition and attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):374-83. doi: 10.1097/00004583-199703000-00016. PMID 9055518
- [Background] Frazier JA, Alaghband-Rad J, Jacobsen L, Lenane MC, Hamburger S, Albus K, Smith A, McKenna K, Rapoport JL. Pubertal development and onset of psychosis in childhood onset schizophrenia. Psychiatry Res. 1997 Apr 18;70(1):1-7. doi: 10.1016/s0165-1781(97)03062-x. PMID 9172272
- [Background] Zahn TP, Jacobsen LK, Gordon CT, McKenna K, Frazier JA, Rapoport JL. Autonomic nervous system markers of psychopathology in childhood-onset schizophrenia. Arch Gen Psychiatry. 1997 Oct;54(10):904-12. doi: 10.1001/archpsyc.1997.01830220020003. PMID 9337769
- [Derived] Loeb FF, Zhou X, Craddock KES, Shora L, Broadnax DD, Gochman P, Clasen LS, Lalonde FM, Berman RA, Berman KF, Rapoport JL, Liu S. Reduced Functional Brain Activation and Connectivity During a Working Memory Task in Childhood-Onset Schizophrenia. J Am Acad Child Adolesc Psychiatry. 2018 Mar;57(3):166-174. doi: 10.1016/j.jaac.2017.12.009. Epub 2017 Dec 28. PMID 29496125